CLINICAL TRIAL: NCT00028821
Title: A Phase I and Pharmacologic Study of 2-Methoxyestradiol in Patients With Advanced Solid Tumors
Brief Title: 2-Methoxyestradiol in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02439; MC0017; U01CA069912 (NIH); CDR0000069137 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Refractory Multiple Myeloma; Stage III Multiple Myeloma; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Multiple Myeloma | interventions — 2-Methoxyestradiol; Mercaptoethanol

ARMS (1):
- Treatment (2-methoxyestradiol) (Experimental): Patients receive oral 2-methoxyestradiol (2-ME) once daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 2-methoxyestradiol; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: 2-methoxyestradiol — Given orally
  Other Names: 2-ME; 2-Methoxy Estradiol; 2ME2; Panzem
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase I trial to study the effectiveness of 2-methoxyestradiol in treating patients who have advanced solid tumors. 2-methoxyestradiol may stop or slow the growth of solid tumors by stopping blood flow to the tumor

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the optimal biologic dose and/or maximum tolerated dose of 2-methoxyestradiol in patients with advanced solid tumors.

II. Determine the qualitative and quantitative toxic effects of this drug in these patients.

III. Determine the pharmacokinetics and metabolism of this drug in these patients.

IV. Determine the biologic changes within the tumor of these patients when treated with this drug.

V. Correlate the pharmacokinetics and toxicity of this drug in these patients. VI. Evaluate the biologic evidence of angiogenesis inhibition in patients receiving this drug.

VII. Correlate genetic polymorphisms in cytochrome P450 and sulfotransferases isoforms with the pharmacokinetics of this drug.

OUTLINE: This is a dose-escalation study.

Patients receive oral 2-methoxyestradiol (2-ME) once daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of 2-ME until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Additional patients are treated at the MTD.

Patients are followed for 3 months.

PROJECTED ACCRUAL: A total of 42-60 patients will be accrued for this study within 19 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor that is clinically unresectable

  * No known standard therapy that is potentially curative or definitely capable of extending life expectancy
  * Patients with multiple myeloma may be enrolled to expansion cohort once the recommended phase II dose is established
* Tumor amenable to serial biopsy
* No bone metastases as only site of disease
* No CNS metastases
* Performance status - ECOG 0-2
* At least 12 weeks
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL
* Bilirubin normal
* AST no greater than 2.5 times upper limit of normal (ULN)
* Creatinine no greater than 1.5 times ULN
* No New York Heart Association class III or IV heart disease
* Adequate oral intake
* No malabsorption syndrome
* No disease of terminal small bowel
* No dysphagia or other condition that would interfere with ability to swallow intact capsules
* No clinical contraindications (e.g., anticoagulant therapy) to biopsy
* No uncontrolled infection
* No seizure disorder
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* More than 4 weeks since prior biologic therapy
* More than 4 weeks since prior immunotherapy
* No concurrent immunotherapy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No concurrent chemotherapy
* No concurrent megestrol
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to more than 25% of bone marrow
* No concurrent radiotherapy
* No prior extensive resection of terminal small bowel
* No prior major resection of the stomach or proximal small bowel
* No other concurrent ancillary investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-01; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) based on the incidence of dose-limiting toxicity (DLT) as assessed by Common Toxicity Criteria (CTC) version 2.0 | 28 days
  Presented primarily in a descriptive fashion.
Number of toxicity incidents as assessed by CTC version 2.0 | Up to 3 months after completion of treatment
  Frequency distributions and other descriptive measures will form the basis of the analysis of these variables.

SECONDARY OUTCOMES:
Biologic activity rate (BAR) | At day 1 and at day 28
  A rate will be calculated by dividing the number of patients with BA by the number of patients treated at the phase II recommended dose level.
Angiogenesis inhibition via an ex vivo angiogenesis assay | At day 1 and at day 28
  The relationship between each marker and dose level will be explored descriptively.
Number of responses | Up to 3 months after completion of treatment
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Erlichman, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States